CLINICAL TRIAL: NCT05764668
Title: Efficacy and Safety of Zihua Wenfei Granules in Treatment of Postinfectious Cough (Wind-cold Invading Lungs Syndrome): a Randomized, Double-blind, Placebo-controlled, Multicenter Phase III Clinical Trial
Brief Title: Efficacy and Safety of Zihua Wenfei Granules in Treatment of Postinfectious Cough (Wind-cold Invading Lungs Syndrome)
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: DoCare Pharmaceutial Technology Co.,Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KCDC-ZHWFZSKLⅢ-2022
Record Dates: First submitted 2023-02-24; First posted 2023-03-13 (Actual); Last update posted 2023-03-13 (Actual); Status verified 2023-02

CONDITIONS: Cough
MeSH Terms: conditions — Cough

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Zihua Wenfei Zhisou Granule (Experimental): Patients in experimental treatment arm were given Zihua Wenfei Zhisou Granule (15 g/bag, one bag at a time, three times/day ). All treatment lasted for 14 days and no other antitussive/decongestant or bronchodilators are given to any patients.
  Interventions: Drug: Zihua Wenfei Zhisou Granule
- Zihua Wenfei Zhisou Granule-matched placebo (Placebo Comparator): Patients in placebo treatment arm were given Zihua Wenfei Zhisou Granule-matched placebo (15 g/bag, one bag at a time, three times/day ). All treatment lasted for 14 days and no other antitussive/decongestant or bronchodilators are given to any patients.
  Placebo does not contain active pharmaceutical ingredients, and its main ingredients are lactose, beta-cyclodextrin, stevioside, and caramel.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Zihua Wenfei Zhisou Granule — 14 daily- doses of Zihua Wenfei Zhisou Granule，one bag at a time (15 g/bag), three times/day
  Arms: Zihua Wenfei Zhisou Granule
Drug: Placebo — 14 daily- doses of placebo，one bag at a time (15 g/bag), three times/day
  Arms: Zihua Wenfei Zhisou Granule-matched placebo

SUMMARY:
Cough is a common symptom of respiratory medicine clinic patients, which has complex etiology and wide-ranging. Cough is usually divided into three categories by time: acute cough, subacute cough and chronic cough. Subacute cough has a 3~8 weeks course of disease. Its main etiology is postinfectious cough, which is mostly secondary to viral infection.The drug in this study is for post-infection cough in subacute cough. After long-term clinical practice, six traditional Chinese medicines, including Aster, Lonicera japonica, Shegan, dried ginger, mango seed and Schizonepeta tenuifolia, were selected to form Zihua Wenfei Zhisou Decoction. This product has the effect of relieving wind, relieving cough, warming the lung and resolving phlegm. It can be used for the cough syndrome caused by Wind-cold invading lungs syndrome. The aim is to evaluate the efficacy and safety of Zihua Wenfei Zhisou Granule in the treatment of postinfection cough (wind-cold lung syndrome) with placebo as a control.

DETAILED DESCRIPTION:
Patients in treatment arm were given Zihua Wenfei Zhisou Granule (15 g/bag, one bag at a time, three times/day). Patients in placebo treatment arm were given Zihua Wenfei Zhisou Granule-matched placebo (15 g/bag, one bag at a time, three times/day). All treatment lasted for 14 days and no other antitussive/decongestant or bronchodilators are given to any patients. After that, there will be a follow-up 14 days after drug withdrawal.

ELIGIBILITY:
Inclusion Criteria:

* When signing the informed consent form, the age is between 18 and 65 years old (including 18 and 65 years old)；
* Diagnosis of postinfectious cough;
* Wind-cold invading lungs syndrome in TCM Zheng;
* Baseline cough visual analogue scale of 60 mm or more;
* Cough duration of 3- 6 weeks;
* Voluntarily provide written and informed consent.

Exclusion Criteria:

* Cough caused by cough variant asthma, upper airway cough syndrome, eosinophilic bronchitis, gastroesophageal reflux cough or any other concomitant conditions;
* Patients with severe pulmonary diseases such as lung cancer, lung tuberculosis, or lung fibrosis;
* After inhaling bronchodilator, patients with FEV1/FVC<70% were excluded;
* Subjects who have taken angiotensin-converting-enzyme inhibitor (ACEI) in the past month;
* Current smokers or recent ex-smokers quitting smoking less than 3 months ago;
* FeNO ≥ 32 ppb or Bronchial provocation test positive (for FeNO and Bronchial provocation test, if the center cannot detect it, it can be detected in other qualified tertiary hospitals);
* Combined with serious cardio-cerebrovascular diseases, malignant tumors, diseases of blood and hematopoietic system, gastrointestinal diseases or other serious or progressive diseases of the system; Or those who are unable to cooperate or unwilling to cooperate due to severe mental illness, severe cognitive impairment, etc;
* Liver and kidney dysfunction: ALT or AST >2 times the upper limit of normal reference value; And/or serum creatinine >1.5 times the upper limit of normal reference value, or eGFR< 60 mL/min/1.73m2;
* White blood cell count < 3.0×109/L or > 10.0×109/L, and/or neutrophil granulocyte > 80%;
* Patients with temperature of 37.3℃ or above;
* Patients taking similar medications in the last one week;
* Have a long history of alcohol or drug abuse;
* Pregnancy or potential pregnancy or lactation;
* Allergic constitution or known to be allergic to any component in tested drug;
* Patients having participated or participating in another trial in last 3 month;
* Patients unsuitable for clinical trials judged by researchers.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 480 (Estimated)
Dates: Start 2022-11-15 (Actual); Primary Completion 2023-11 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
Cough relief rate | day 14
  Cough relief refers to a 50% or more reduction in cough VAS score

SECONDARY OUTCOMES:
Complete remission rate of cough | day 14
  Complete remission of cough refers to cough VAS score<17 mm
Time to cough relief | day 14
  Time to cough relief
Complete remission time of cough | day 14
  Complete remission time of cough
Change from baseline in Cough Evaluation Test (CET) value | day 0、day 7、day 14
  Change from baseline in Cough Evaluation Test (CET) value
Change from baseline in visual analogue scale (VAS) value | day 0、day 7、day 14
  The visual analogue scale (VAS) is a 100 mm scale, with a minimum value of 0 mm and a maximum value of 100 mm. 0 mm means that the cough is not troubled at all, and 100 mm means that the cough is the most troubled.
Change from baseline in TCM syndrome score | day 0、day 7、day 14
  Change from baseline in TCM syndrome score
Change from baseline in Leicester Cough Questionnaire (LCQ) score | day 0、day 14、day 28
  The LCQ comprises 19 items and takes 5 to 10 minutes to complete. The LCQ is a validated QoL measurement tool for non-specific cough and assesses the impact of cough on various aspects of life, including emotions, sleeping behaviour, work and relationships. It contains 19 items which are divided over 3 domains: physical (8 items), psychological (7 items) and social (4 items), with a 7-point Likert response scale.

CONTACTS AND LOCATIONS:
Locations (1):
- West China Hospital of Sichuan University, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No